CLINICAL TRIAL: NCT03586024
Title: Phase I/II Study of Pembrolizumab in Patients With Relapsed or Refractory Extranodal NK/T- Cell Lymphoma (ENKTL), Nasal Type and EBV-associated Diffuse Large B Cell Lymphomas (EBV-DLBCL)
Brief Title: Pembrolizumab in Relapsed or Refractory Extranodal NK/T- Cell Lymphoma, Nasal Type and EBV-associated Diffuse Large B Cell Lymphomas
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: poor accrual
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 54417
Record Dates: First submitted 2018-07-03; First posted 2018-07-13 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-04

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: 2 parallel cohort
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort 1 (Experimental): cohort 1: NK/T-cell lymphoma;
  Interventions: Drug: Pembrolizumab
- Cohort 2 (Experimental): EBV-associated diffuse large B cell lymphomas
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — dose of pembrolizumab will be 200 mg IV every 3 weeks

SUMMARY:
To determine the safety and efficacy (overall response rate) of pembrolizumab in patients with relapsed or refractory ENKTL, and EBV-DLBCL

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the trial.
* Be ≥ 18 years of age on day of signing informed consent.
* Have measurable disease based on defined as at least one lesion that can be accurately measured in at least two dimensions with a spiral CT scan, PET/CT scan, or MRI. Minimum measurement of >1.5 cm in longest diameter by > 1.0 cm in short axis.
* Have a performance status of 0 or 1 on the ECOG Performance Scale.
* Demonstrate adequate organ function, all screening labs should be performed within 10 business days of treatment initiation with the exception of beta-HCG (72 hours), if applicable.
* Female subject of childbearing potential should have a negative serum pregnancy within 72 hours prior to receiving the first dose of study medication.
* Male subjects of childbearing potential (Section 5.7.1) must agree to use an adequate method of contraception as outlined in Section 5.7.1- Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy within 4 weeks of first dose of treatment or used an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has a known history of active TB (Bacillus Tuberculosis)
* Hypersensitivity to pembrolizumab or any of its excipients.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.
* Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
* Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Has undergone prior allogenic hematopoietic stem cell transplantation.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has known history of, or any evidence of active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2020-08-19 (Actual); Study Completion 2020-08-19 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Schuster, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No